CLINICAL TRIAL: NCT04700696
Title: Enhancing Permanency in Children and Families
Acronym: EPIC
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ohio State University (Other)
Collaborators: Children's Bureau - Administration for Children and Families (Other); Pickaway County Job and Family Services (Unknown); Fairfield County Job and Family Services (Unknown); Integrated Services for Behavioral Health (ISBH) (Unknown); Ohio Guidestone (Unknown); Fairfield County Juvenile Court (Unknown); Pickaway County Juvenile Court (Unknown)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 90CU0083-01-00
Record Dates: First submitted 2020-11-10; First posted 2021-01-08 (Actual); Last update posted 2024-01-23 (Actual); Status verified 2022-09

CONDITIONS: Substance Abuse; Substance Use; Child Abuse; Neglect, Child
Keywords: Substance Abuse; Child welfare; Child abuse and neglect
MeSH Terms: conditions — Substance-Related Disorders | interventions — Dosage Forms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- EPIC Participants (Experimental): EPIC participants are 1) matched with trained peer recovery supporters with lived experience related to child welfare and substance EPIC participants are also incentivized to participate in 2) family treatment drug court (FTDC), with medications for opioid use disorders (MOUD); and 3) home-based parenting supports based on the Nurturing Parenting Program.
  Interventions: Behavioral: Peer Recovery Support; Behavioral: Family Treatment Drug Court with Medications for Opioid Use Disorders (MOUD); Behavioral: Relational Skill Building based on the Nurturing Parenting Program (NPP)
- Ohio Sobriety Treatment And Reducing Trauma (START) participants (Active Comparator): Adapted from the evidence-based national START model (Sobriety Treatment and Recovery Teams) this intervention matches child welfare parents in need of addiction services to caseworker and family peer mentor (FPM) dyads for intensive case management services.
  Interventions: Behavioral: Peer Recovery Support
- Treatment as usual (TAU) (No Intervention): Treatment as usual includes home visits by the assigned caseworker, referrals to SUD assessment/treatment, family group decision making, and (non-incentivized) referral to FTDC.

INTERVENTIONS:
Behavioral: Peer Recovery Support — Weekly visits with peer who has lived experience related to child welfare and addiction
  Arms: EPIC Participants; Ohio Sobriety Treatment And Reducing Trauma (START) participants
Behavioral: Family Treatment Drug Court with Medications for Opioid Use Disorders (MOUD) — Incentivized to participate in Family Treatment Drug Court with option for Medications for Opioid Use Disorders (MOUD)
  Arms: EPIC Participants
Behavioral: Relational Skill Building based on the Nurturing Parenting Program (NPP) — Home-based parenting support
  Arms: EPIC Participants

SUMMARY:
The Enhancing Permanency in Children and Families (EPIC) program is a collaborative effort between the Ohio State University College of Social Work, two county offices of the Ohio Department of Job and Family Services, two juvenile courts and local behavioral health agencies. The goal of EPIC is to use three evidence-based and evidence-informed practices to reduce abusive and neglectful parenting, reduce addiction severity in parents, and improve permanency outcomes for families involved with the child welfare system due to substance abuse.

DETAILED DESCRIPTION:
Funded by the federal Regional Partnership Grant (RPG) Program, the Enhancing Permanency in Children and Families (EPIC) is a partnership between child welfare, juvenile count and behavioral health to holistically address substance misuse and associated parenting needs of child welfare-involved families. The overall goals and objectives of the intervention are to 1) Increase timely access to services among substances abusing parents involved in the child welfare system in Fairfield and Pickaway counties, 2.Enhance child safety and improve permanency and 3. increase child, parent, and caregiver well-being.

Eligible participants are matched with peer recovery supporters who mentor parents through the process. Parents are also referred to Family Treatment Drug Court (FTDC) with the option to receive Medications for Opioid Use Disorders (MOUD), and lastly when children are placed at home with parents or with kinship caregivers, relational skill building services that include financial assistance for child care, respite and transportation services. EPIC participants receive substance abuse and behavioral health treatment services through local providers including from two partner agencies: Integrated Services for Behavioral Health and Ohio Guidestone.

Data collection: Participating parents complete a pretest at baseline and up to 5 post-tests at 6 month intervals. Parents complete questions related to themselves (e.g. Addiction Severity Index, CES-D) and for one focal child (e.g. CBCL).

To evaluate EPIC, a quasi-experimental design will be employed through a two-stage sampling procedure. This design provides the ability to assess (1) the effects of EPIC on access to services for the families in the two intervention counties, and (2) the independent effects of additional services provided under EPIC that may be over and above Ohio START (an intervention administered through the Public Children Services Association of Ohio) and treatment as usual (TAU). In the first stage, two comparison counties will be identified for each of the two intervention counties. One comparison county will be part of the Ohio START program while the second will be a county that has no major interventions to address substance use among child welfare families. Counties are matched based on child population size, rate of child protective services referrals, percent of naloxone administrations per adult population, percent white, percent poverty, child welfare tax levy, and to the extent possible, behavioral health service availability. During the second stage, EPIC families are matched with substance using families in each of the comparison counties.

Parents may consent to one or all three components of EPIC based on the specific needs of each family, however all parents receive intensive case management services, including frequent home visits from caseworkers and peer recovery supporters.

ELIGIBILITY:
Inclusion Criteria:

* Child welfare involvement
* Substance use is primary reason for child welfare involvement (a score or 3 or more on UNCOPE assessment or a positive drug screen)

Exclusion Criteria:

* Possible substance use, though not primary reason for child welfare involvement
* incarcerated parents (may enroll after release)

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 117 (Actual)
Dates: Start 2017-10-01 (Actual); Primary Completion 2023-07-01 (Actual); Study Completion 2023-09-30 (Actual)

PRIMARY OUTCOMES:
Time from opening of child welfare case to SUD screening | Within 30 days of program entry
  Measures: 1) Child welfare case open date; 2) UNCOPE assessment screening date Analyses: We will use T-tests to estimate mean differences in the length of time from entry into child welfare and SUD screening for EPIC participants in comparison to Ohio START and treatment as usual.
Time from opening of child welfare case to trauma screening | Within 30 days of program entry
  Measures: Time from opening of child welfare case to trauma screening will be estimated using 1) child welfare case open date; 2) ACEs assessment date for adults or 3) CTAC assessment dates for children.
  Analyses: We will use t-tests to estimate mean differences in the length of time from entry into child welfare and trauma screening for EPIC participants in comparison to Ohio START and treatment as usual.
Change in wait time between referral to addiction treatment services and initiation of services. | Within 30 days of entering child welfare system
  Measures: Change in wait time will be estimated using service referral and service initiation dates.
  Analyses: We will use t-tests to estimate mean differences in the length of time between SUD treatment service referral and service initiation for EPIC participants in comparison to Ohio START and treatment as usual.
Change in addiction severity among participating parents | At program entry and again at program completion. An average of I year
  Measures: Addiction Severity Index-Self Report (ASI-SR) Analyses: A paired sample t-test will be conducted to examine the change in mean scores on the ASI-SR pre and post participation.
Change in resilience in children | At program entry and again at program completion. An average of I year
  Measures: Resilience in children is measured using the Protective Factors Survey (PFS) Analyses: A paired sample t-test will be conducted to examine change in mean scores on the PFS pre and post participation.
Change in child behavior | At program entry and again at program completion. An average of I year
  Measures: The Child Behavior Checklist (CBCL) is used to screen for emotional, behavioral and social problems among children.
  Analyses: A paired sample t-test will be conducted to examine change in mean scores on the CBCL pre and post participation.
Change length of stay in out-of-home placement for children in EPIC program compared to substance-affected families not receiving EPIC. | Through program completion, an average of 1 year.
  Data source: Statewide Automated Child Welfare Information System (SACWIS), obtained twice a year through study completion.
  Measures: Length of stay in out-of-home placement will be operationalized using placement dates obtained in SACWIS.
  Analyses: Survival analysis will be utilized to study outcome measures (e.g., length of stay in out-of-home placement) Due to the likelihood of censored measures when we have families who are still involved in the child welfare system, particularly for families who enter the system near the end of the study period, we will use survival analysis to estimate treatment effects on length of stay in out of home placement in comparison to Ohio START and treatment as usual families.
Change in reunification among families involved in EPIC compared to substance-affected families not receiving EPIC. | Through program completion, an average of 1 year.
  Data source: Statewide Automated Child Welfare Information System (SACWIS), obtained twice a year through study completion.
  Analyses: Logistic regression will be used to estimate treatment effects on in comparison to Ohio START and treatment as usual.
Change in subsequent child welfare involvement among parents receiving EPIC compared to substance-affected families not receiving EPIC | Through completion of 5 year study. For participants, up to 4 years following program participation, depending on time of enrollment
  Data source: Statewide Automated Child Welfare Information System (SACWIS), obtained twice a year through study completion.
  Measures: Subsequent child welfare entry (yes/no) is measured using re-entry dates in SACWIS.
  Analyses: Logistic regressions will be used to estimate treatment effects on subsequent child welfare involvement in comparison to Ohio START and treatment as usual.

CONTACTS AND LOCATIONS:
Overall Officials: Bridget Freisthler, Principal Investigator — Ohio State University
Locations (1):
- The Ohio State University, Columbus, Ohio, United States

IPD SHARING:
Plan to Share IPD: Yes
Datasets will be be stripped of identifying information prior to construction. Specifically, parents (along with one focal child) will be identified with a case and individual identification numbers. No names, addresses, telephone numbers, fax numbers, email addresses, social security numbers, child welfare records, etc. will be retained. We will only share data with external investigators when a data use agreement (DUA) is executed between the Ohio State University and the requester's institution. The DUA will specify the requested data elements (each of which must be justified), the specific research question and the timeline for the project. These data will be made available in Fall, 2023 by the PI.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: Fall 2023
Access Criteria: With permission via study website
URL: https://u.osu.edu/epic/

REFERENCES:
- [Derived] Shockley McCarthy K, Price Wolf J, Dellor E. Promoting permanency in families with parental substance misuse: lessons from a process evaluation of a multi-system program. BMC Public Health. 2022 Dec 3;22(1):2261. doi: 10.1186/s12889-022-14528-4. PMID 36463173
- [Derived] Freisthler B, Maguire-Jack K, Yoon S, Dellor E, Wolf JP. Enhancing Permanency in Children and Families (EPIC): a child welfare intervention for parental substance abuse. BMC Public Health. 2021 Apr 23;21(1):780. doi: 10.1186/s12889-021-10668-1. PMID 33892671
- See also: Study website — https://u.osu.edu/epic/